CLINICAL TRIAL: NCT05199012
Title: Safety and Efficacy of Oral Supplementation With a Black Pepper Extract in Apparently Healthy Men and Women
Brief Title: Oral Supplementation With a Black Pepper Extract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Applied Health Sciences, LLC (Industry)
Collaborators: Brightseed, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: #21-CAHS-103
Record Dates: First submitted 2021-12-17; First posted 2022-01-20 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Waist Circumference; Triglycerides; Appetite; Inflammation; Lipids
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo is maltodextrin, delivered as 2 capsules.
  Interventions: Dietary Supplement: Black pepper extract
- Active (Active Comparator): The active comparator is black pepper extract, delivered as 2 capsules.
  Interventions: Dietary Supplement: Black pepper extract

INTERVENTIONS:
Dietary Supplement: Black pepper extract — Subjects will be randomized to receive either the placebo or active (black pepper extract) in a 1:1

SUMMARY:
This study is a randomized, placebo-controlled, double-blind, two-arm trial of N=94 apparently healthy men and women to be recruited at a single investigational center in Northeast Ohio. Subjects will attend three study visits. During Visit 1, subjects will be screened for participation (i.e., medical history, physical exam, routine blood work, background baseline diet). Over the next 12 weeks, subjects will attend Visits 2 (baseline) and 3 (week 12), wherein assessments of body weight, waist circumference, urinary ketones, serum glucose, insulin, liver enzymes as well as other biomarkers of metabolic health, quality of life (SF-36 questionnaire), and various visual analog scales (VAS) for appetite, satiety, and cravings will be made.

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntary signed and dated informed consent.
* Be in good health as determined by medical history and routine blood chemistries.
* Age between the ages of 21 and 65 (inclusive).
* Body Mass Index of 25-34.99 (inclusive).
* Body weight of at least 120 pounds.
* Normotensive (seated, resting systolic blood pressure <140 mm Hg and diastolic blood pressure < 90 mm Hg. If the first measurement is slightly elevated above these limits, the subject will be given a brief (5 minute) rest period, and two more measurements will be taken. The average of all three measurements will be used to determine eligibility.
* Normal seated, resting heart rate (<90 per minute).
* Willing to duplicate their previous 24-hour diet, refrain from caffeine for 12 hr, abstain from exercise for 24 hr, and fast for 10 hours prior to each laboratory visit.

Exclusion Criteria:

* History of unstable or new-onset cardiovascular or cardiorespiratory disease.
* Individuals diagnosed with diabetes or other endocrine disorder.
* Fasting blood sugar of > 126 mg/dL OR HgA1c of > 6.5%.
* History of use of medications or dietary supplements known to affect glycemia or insulinemia.
* Current use of amiodarone, anti-retroviral agents, corticosteroids, methotrexate, tamoxifen, valproate, amitriptyline (Elavil), codeine, desipramine (Norpramin), flecainide (Tambocor), haloperidol (Haldol), imipramine (Tofranil), metoprolol (Lopressor, Toprol XL), ondansetron (Zofran), paroxetine (Paxil), risperidone (Risperdal), tramadol (Ultram), venlafaxine (Effexor), cyclosporine, lithium, chlorzoxazone, theophylline, and bufuralol, cyclophosphamide, ifosfamide, barbiturates, bromobenzene, lovastatin (Mevacor), ketoconazole (Nizoral), itraconazole (Sporanox), fexofenadine (Allegra), triazolam (Halcion), glimepiride (Amaryl), glyburide (DiaBeta, Glynase PresTab, Micronase), insulin, pioglitazone (Actos), rosiglitazone (Avandia), etoposide, paclitaxel, vinblastine, vincristine, vindesine, amprenavir, indinavir, nelfinavir, saquinavir, cimetidine, ranitidine, diltiazem, verapamil, digoxin, erythromycin, cisapride (Propulsid),, loperamide (Imodium), quinidine, aspirin, clopidogrel (Plavix), dalteparin (Fragmin), enoxaparin (Lovenox), heparin, ticlopidine (Ticlid), warfarin (Coumadin), nevirapine, Pentobarbital (Nembutal), Phenytoin (Dilantin), Propranolol (Inderal), Rifampin, Amoxicillin (Amoxil, Trimox), Carbamazepine (Tegretol), Cefotaxime (Claforan), midazolam, diclofenac.
* History of hyperparathyroidism or an untreated thyroid disease.
* History of nephrotic syndrome or renal disease.
* History of alcohol abuse within the past year.
* History of malignancy in the previous 5 years except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin).
* Prior gastrointestinal bypass surgery (Lapband), etc.
* Other known gastrointestinal or metabolic diseases that might impact nutrient absorption or metabolism, e.g., short bowel syndrome, diarrheal illnesses, history of colon resection, gastro paresis, Inborn-Errors-of-Metabolism (such as PKU).
* Chronic inflammatory condition or autoimmune disease (e.g., rheumatoid arthritis, hepatitis, Crohn's disease, ulcerative colitis, Lupus, HIV/AIDS, etc.).
* Female subjects who are pregnant, trying to become pregnant, or lactating. Women who participate in this study must agree to the use of contraception for the duration of the study and any woman that is sexually active will have to have a negative pregnancy test prior to enrolling. Women of childbearing age (any woman prior to menopause or surgically sterilized) regardless of their use of contraception will be provided a urine pregnancy test kit at their screening visit and take the test in private using the female lavatory after signing an informed consent.
* Known sensitivity to any ingredient in the test formulations as listed in the Certificates-of- Analysis.
* Currently participating in another research study with an investigational product or have been in another research study in the past 30 days.
* Any other diseases or conditions that, in the opinion of the medical staff, could confound the primary endpoints or place the subject at increased risk of harm if they were to participate.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
waist circumference | Change from baseline to week 12
  measurement of waist circumference in centimeters
triglycerides | Change from baseline to week 12
  measurement of triglycerides in blood

SECONDARY OUTCOMES:
urinary ketones | Change from baseline to week 12
  ketone concentration in urine
plasma free fatty acids | Change from baseline to week 12
  concentration of free fatty acids in plasma
body weight | Change from baseline to week 12
  body weight measurement in kg
Body mass index | Change from baseline to week 12
  body mass index (body weight relative to height)
liver enzymes | Change from baseline to week 12
  fasting levels of ALT and AST measured in international units per liter (IU/L)

OTHER OUTCOMES:
Appetite | Change from baseline to week 12
  appetite as measured with a 10 cm anchored visual analogue scale, where higher values represent greater cravings.
Satiety | Change from baseline to week 12
  satiety as measured with a 10 cm anchored visual analogue scale, where higher values represent greater satiety.
Cravings | Change from baseline to week 12
  cravings as measured with a 10 cm anchored visual analogue scale, where higher values represent greater cravings.
Short Form Health Survey (SF-36) | Chnage from baseline to week 12
  health status as measured with the SF-36 questionnaire, where scores range from 0 to 100, and higher values represent better health status.

CONTACTS AND LOCATIONS:
Locations (1):
- The Center for Applied Health Sciences, Canfield, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided